CLINICAL TRIAL: NCT05590169
Title: Comparison of Effects of Telerehabilitation-based Individual and Group Exercises on Functional Capacity in Patients with Cystic Fibrosis
Brief Title: Effects of Telerehabilitation-based Exercises in Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Bilgi University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Cigdem Emirza, Research Assistant, Istanbul Bilgi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05112022/96
Record Dates: First submitted 2022-10-16; First posted 2022-10-21 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2024-02

CONDITIONS: Cystic Fibrosis; Exercise; Telerehabilitation; Exercise Capacity
Keywords: physiotherapy; cystic fibrosis; randomized controlled trial; telerehabilitation
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group I (Experimental): They will be included in exercise training as a group (three or four participants) with telerehabilitation (via Zoom application) for eight weeks. Exercise program includes: (F) 3 times a week, (I) at 60-70% of the maximum heart rate, (T): breathing, stretching, aerobic, plyometric, balance exercises, (T) 30 minutes each session, a total of 8 week. During the exercise sessions, the heart rate will be monitored via a Polar Unite Fitness Watch, and the oxygen saturations will be monitored with a pulse oximeter.
  Interventions: Other: Exercise training
- Group 2 (Experimental): They will be individually included in exercise training with (via Zoom application) for eight weeks. Exercise program includes: (F) 3 times a week, (I) at 60-70% of the maximum heart rate, (T): breathing, stretching, aerobic, plyometric, balance exercises, (T) 30 minutes each session, a total of 8 week. During the exercise sessions, the heart rate will be monitored via a Polar Unite Fitness Watch, and the oxygen saturations will be monitored with a pulse oximeter.
  Interventions: Other: Exercise training
- Group 3 (No Intervention): They will continue their routine treatment (medical treatment, airway cleaning techniques, physical activity counseling).

INTERVENTIONS:
Other: Exercise training — Group 1: Group exercises via Zoom application Group 2: Individual exercises via Zoom application Group 3: Routine treatment
  Other Names: Telerehabilitation-based exercise
  Arms: Group 2; Group I

SUMMARY:
Pulmonary rehabilitation programs are an important part of lifelong therapy in the treatment of patients with cystic fibrosis. Although the possible benefits of exercise are known, physical activity levels and participation in exercise are low in patients with cystic fibrosis. There are barriers such as lack of time, demoralization, lack of motivation, and transportation problems. Although group exercises are an approach that increases participation and motivation, it is not considered a very suitable method because it increases the risk of cross infection in patients with cystic fibrosis when performed face-to-face. Telerehabilitation programs, which are increasingly used in chronic respiratory diseases, show similar results with clinical rehabilitation programs. Telerehabilitation programs, the effects of which have been examined in different disease groups in recent years, on patients with cystic fibrosis are limited in the literature. Group exercises that can be given with the telerehabilitation method may be a good approach for patients with cystic fibrosis, eliminating possible infection transmission.

The goal of this interventional clinical trial is to compare of effects of telerehabilitation based individual and group exercises on functional exercise capacity, muscle strength, respiratory functions, balance, anaerobic power, quality of life, and adherence in children with cystic fibrosis. The main question it aims to answer are:

• Is there a difference between functional exercise capacity, muscle strength, respiratory functions, balance, anaerobic performance, quality of life and compliance with treatment between telerehabilitation based group exercises and telerehabilitation based individual exercises in patients with cystic fibrosis?

Participants will be randomized into three groups:

Group 1: They will be divided into groups of four and included in the exercise training for eight weeks with telerehabilitation.

Group 2: They will be individually included in exercise training with telerehabilitation for eight weeks.

Group 3 (control group): They will continue their routine treatment (medical treatment, airway cleaning techniques, physical activity counseling).

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with cystic fibrosis
* Being between the ages of 8-18
* Having a device for video calls (phone, computer, tablet, etc.)

Exclusion Criteria:

* Severe airway obstruction (FEV1 (%, predicted) <40%)
* Pulmonary exacerbation/hospitalization in the last four weeks
* History of lung transplant
* Orthopedic problems that limit exercise
* Those who had a change in their medical treatment during the study

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2023-05-20 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Functional exercise capacity | 0-8 weeks
  Six-minute walking test: Before the test, oxygen saturation, heart rate, blood pressure, dyspnea and fatigue measurements are recorded. The patient walks for six minutes as fast as they can walk on the ground for at least 30 meters. The walking distance is recorded in meters. If the patient stops during the test, the total time he stopped, the number of times he stopped is recorded. After the test, the evaluations made before the test are repeated.
Functional exercise capacity | 0-8 weeks
  Modified shuttle walking test: It is a maximal test performed by adjusting walking speed with pre-recorded signals. Before the test, oxygen saturation, heart rate and blood pressure, dyspnea and fatigue will be recorded. The patient walks between two 10-meter points. Walking speed is increased every minute. The test is terminated when the required speed cannot be maintained or the speed cannot be followed. At the end of the test, the measurements are repeated.

SECONDARY OUTCOMES:
Muscle strength | 0-8 weeks
  For the peripheral muscle strength, the strength and grip strength of the knee extensor, hip flexor and abductor muscles in the lower extremity, and the elbow flexor, shoulder flexor and abductor muscles in the upper extremity will be examined. Measurement of muscle strength will be made with a Lafayette manual muscle tester, measurement of grip strength will be made with a Jamar hydraulic hand dynamometer. Evaluations will be made with the patient in a sitting position with back support. Evaluation of muscle strength will be done by evaluating the right and left extremities, and the grip strength will be repeated three times separately for the dominant hand and the non-dominant hand.
Spirometric measurements | 0-8 weeks
  The measured and predictive (%) values of FEV1, forced vital capacity (FVC), FEV1/FVC ratio, peak expiratory flow (PEF) will be recorded from the results of the pulmonary function test performed in accordance with the American Thoracic Society/European Respiratory Society guidelines.
Balance | 0-8 weeks
  Timed up and go test will use for balance assessment. The test, which starts with sitting in a chair, ends with walking a distance of three meters, turning and sitting on the chair again. The test completion time is recorded in seconds.
Anaerobic performance | 0-8 weeks
  The anaerobic performance of the patients will be evaluated with the vertical jump test. The vertical jump test is an indicator of lower extremity explosive strength. When the patient jumps as high as possible, the distance achieved by the jump is recorded in meters. The test is repeated three times and the best performance is recorded.
Health-related quality of life by questionnaire | 0-8 weeks
  The Pediatric Quality of Life Inventory (PedsQL) developed by Varni et al. will be used to evaluate the quality of life of the patients. The scale consists of 23 items in total. Eight of these items question physical, five emotional, five social, and five school functionality. The total score is calculated by scoring each item on a five-point Likert scale (0-4). The higher the score, the better the health-related quality of life.
Adherence rate | When the exercise training is over (after eight weeks)
  An exercise diary will be given to monitor the patients' daily routine physiotherapy (airway cleaning techniques, physical activity, etc.). Sessions will be logged by patients and their families. At the end of the treatment, the continuity of the routine treatment will be calculated as % with the equation "routine treatment sessions x 100/total days". A record of participation in telerehabilitation-based supervised exercise sessions will be recorded by the physiotherapist. When the training is over, the adherence rate will be calculated as % with the equation "exercise sessionsx100/24".

CONTACTS AND LOCATIONS:
Overall Officials: Goksen Kuran Aslan, PT, phD, Study Director — Istanbul University - Cerrahpasa
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul University-Cerrahpasa, Istanbul, Istanbul
  - Istanbul Bilgi University, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen JJ, Cooper DM, Haddad F, Sladkey A, Nussbaum E, Radom-Aizik S. Tele-Exercise as a Promising Tool to Promote Exercise in Children With Cystic Fibrosis. Front Public Health. 2018 Sep 28;6:269. doi: 10.3389/fpubh.2018.00269. eCollection 2018. PMID 30324099
- [Background] Stanford G, Daniels T, Brown C, Ferguson K, Prasad A, Agent P, Gates A, Morrison L. Role of the Physical Therapist in Cystic Fibrosis Care. Phys Ther. 2022 Dec 30;103(1):pzac136. doi: 10.1093/ptj/pzac136. PMID 36193006
- [Background] Cox NS, Dal Corso S, Hansen H, McDonald CF, Hill CJ, Zanaboni P, Alison JA, O'Halloran P, Macdonald H, Holland AE. Telerehabilitation for chronic respiratory disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013040. doi: 10.1002/14651858.CD013040.pub2. PMID 33511633